CLINICAL TRIAL: NCT04926259
Title: Tau PET Imaging With 18F-T807(AV1451) in Neurodegenerative Disorders
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Shaobo Yao, PhD, Director of Nuclear Medicine Department, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRCTA, ECFAH of FMU [2021]129
Record Dates: First submitted 2021-06-07; First posted 2021-06-15 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Neurodegenerative Disorders
MeSH Terms: conditions — Neurodegenerative Diseases | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-T807, PET/CT (Experimental): PET/CT perform after injecting 18F-T807
  Interventions: Drug: 18F-T807

INTERVENTIONS:
Drug: 18F-T807 — Intravenous injection of one dose of 10mCi (370MBq, ±5%) 18F-T807. Each subject receive a single intravenous injection of 18F-T807, and undergo PET/CT imaging within the specificed time.

SUMMARY:
Alzheimer's disease, Parkinson's disease, and Huntington's disease are common neurodegenerative diseases. Tau is a microtubule-associated protein, and aggregated tau resulting from hyperphosphorylation is a pathological feature of a group of neurodegenerative diseases known as tauopathies. The 18F-T807 (AV1451) molecular probe is a novel molecularly targeted imaging agent that exhibits high affinity and good selectivity for tau.

DETAILED DESCRIPTION:
In this study, 18F-T807 (AV1451) molecular probe PET/CT was used to monitor the regional distribution and the degree of deposition in patients with neurodegenerative diseases, and compared with clinical symptoms to evaluate its value in the early differential diagnosis of neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients or their families complain of significant memory impairment;
* Objective memory impairment (e.g., tests of article identification, recall, delayed memory);
* Be able to obtain complete diagnosis and treatment records and be able to carry out long-term follow-up;
* Signed written consent.

Exclusion Criteria:

* Psychiatric disorders: including anxiety disorder, affective disorder, severe psychosis, or drug-induced psychosis;
* Pregnancy or lactation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
standardized uptake value ratio (SUVR) | From right after tracer injection to 2-hours post-injection
  the ratio of radioactivity in a cerebral region to that in the cerebellum as a reference
Aβ42 in CSF | Within 2 hours prior to tracer injection
  Aβ42 (amyloid beta isoform 42) is significantly lower in the cerebrospinal fluid of patients with neurodegenerative diseases and is one of the biomarkers used clinically to diagnose neurodegenerative diseases
t-tau in CSF | Within 2 hours prior to tracer injection
  t-tau (total tau) is significantly increased in the cerebrospinal fluid of patients with neurodegeneration and is one of the biomarkers used clinically to diagnose neurodegeneration
p-tau in CSF | Within 2 hours prior to tracer injection
  p-tau (tau phosphorylated at Thr-181) is significantly increased in the cerebrospinal fluid of patients with neurodegeneration and is one of the biomarkers used clinically to diagnose neurodegeneration
NfL in CSF | Within 2 hours prior to tracer injection
  NfL (neurofilament light chain) is significantly increased in the cerebrospinal fluid of patients with neurodegeneration and is one of the biomarkers used clinically to diagnose neurodegeneration
NfL in the blood | Within 2 hours prior to tracer injection
  NfL is significantly increased in the blood of patients with neurodegeneration and is one of the biomarkers used clinically to diagnose neurodegeneration

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No